CLINICAL TRIAL: NCT02983188
Title: A Double-blind, Randomized, Placebo-controlled Trial of Berberine as an Adjuvant to Treat Antipsychotic-induced Metabolic Syndrome in Patients With Schizophrenia Spectrum Disorders
Brief Title: Berberine as Adjuvant Treatment for Schizophrenia Patients
Acronym: BER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Kowloon Hospital, Hong Kong (Other); Castle Peak Hospital (Other Government); Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, Associate Director (Clinical Affairs), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 17-020
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Metabolic Syndrome x
Keywords: Schizophrenia; Berberine; Metabolic Syndrome; Chinese medicine; Herbal medicine
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Metabolic Syndrome | interventions — Berberine; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine (Active Comparator): Patients will receive berberine pills in additional to current atypical antipsychotic agents
  Interventions: Drug: Berberine; Drug: Antipsychotic Agents
- Placebo (Placebo Comparator): Patients will receive placebos pills in additional to current atypical antipsychotic agents
  Interventions: Drug: Placebos; Drug: Antipsychotic Agents

INTERVENTIONS:
Drug: Berberine — Berberine tablets, 0.3g every time, two times daily
  Arms: Berberine
Drug: Placebos — Placebo tablets, 0.3g every time, two times daily
  Other Names: Placebo
  Arms: Placebo
Drug: Antipsychotic Agents — Antipsychotic agents prescribed at the discretion of the patients' psychiatrists with respect to patients' conditions. Concomitant use of other psychotropic drugs, including antidepressants, anxiolytics, and mood stabilizers for mood disorders, benzodiazepines and non-benzodiazepines for insomnia, and anticholinergics for extrapyramidal symptoms, was allowed as usual. For those who were under anti-hyperlipidemic, antihypertensive and anti-diabetic treatment, they were allowed to continue their current medications throughout the study.

SUMMARY:
One double-blind, randomized, placebo-controlled trial is designed to examine whether berberine added to current antipsychotic drugs could produce significantly greater efficacy in reducing atypical antipsychotic-induced metabolic syndrome. To achieve this objective, 120 patients with schizophrenia spectrum disorders (SSD) who have developed metabolic syndrome will be recruited and randomly assigned to receive additional treatment with placebo (n = 60) or berberine (n = 60, 0.6 g/day, 0.3 g, b.i.d.) for 12 weeks. The primary outcome is changes in net weight gain; other outcomes include body mass index (BMI), waist circumference (WC), blood pressure, triglycerides (TG), total cholesterol, high-density lipoprotein (HDL), and low-density lipoprotein (LDL), fasting glucose, glycated haemoglobin (HbA1c).

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that affects about 1% of the worldwide population. Most patients develop a chronic course with frequent relapses and exacerbation of symptoms and required to have long-term treatment. Although antipsychotic therapy is the mainstay of the management of schizophrenia, the treatment outcomes are often unsatisfactory, largely due to adverse drug reactions. Metabolic syndrome is a highly prevalent side effect incurred in antipsychotic therapy, with a prevalence of 35% in patients with severe mental illness in Hong Kong. No effective therapies are available in treating antipsychotic-induced metabolic syndrome, although some antidiabetic medications may have limited benefits in controlling weight gain and increased glucose level.

Berberine is a natural plant alkaloid isolated from the Chinese herb, Coptis chinensis (Huang-Lian), which is traditionally used for diarrhea caused by bacterial and viral infections in clinical practice. Several lines of evidence suggest that berberine has body weight-lowering, anti-diabetic, and anti-hyperlipidemic effects. One recent study has further shown that the addition of berberine significantly prevented olanzapine (OLZ)-Induced weight gain in rats and modulated the expression of multiple key genes that control energy expenditure.

In addition to the peripheral effects, berberine also broadly modulates brain biogenic amines and related receptors that are involved in the pathogenesis of antipsychotic-induced metabolic syndrome. This suggests that it may be suitable for the treatment of antipsychotic-induced metabolic disturbance.

Over the past decade, a number of studies have demonstrated comparable efficacy of berberine as mono- and combination therapy in reducing metabolic symptoms, without serious side effect. The efficacy of berberine also has been well confirmed in patients with gastrointestinal, liver, heart, and ovary disease as well as in renal-transplant recipients and healthy volunteers. It is well tolerated and only minor digestive reactions were observed, mainly nausea, diarrhea, constipation, abdominal distension and pain.

The results obtained from the clinical and animal studies of the group strongly suggest the promising effects of berberine against OLZ-induced weight gain, without changing pharmacokinetic and pharmacodynamics profile of OLZ at peripheral and central levels. This warrants further evaluation in a larger randomized controlled trial.

The working hypothesis of the proposed study is that berberine as an adjuvant can control weight gain and other metabolic symptoms associated with antipsychotic therapy. To test this hypothesis, a 12-week, double-blind, randomized, placebo-controlled trial will be conducted in patients with schizophrenia spectrum disorders (SSD) to determine whether berberine adjunctive treatment could limit weight gain and improve other anthropometric and metabolic measures in patients with SSD who have developed metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of SSD, including schizophrenia, schizoaffective disorder, schizophreniform disorder, and psychotic disorder not otherwise specified according to the Classification of Mental and Behavior Disorders (10th version);
* have been under atypical antipsychotic treatment for at least 3 months and current conditions are stable, indicated by no difficulty to communicate with investigators and give informed consent; and
* have developed metabolic syndrome according to the International Diabetes Federation criteria for metabolic syndrome in Asian/Chinese population.

Exclusion Criteria:

* serious comorbid gastrointestinal or other unstable medical conditions;
* have suicidal ideas or attempts or aggressive behavior;
* have a history of alcohol abuse in the past 3 months;
* have a history of drug abuse in past 3 months;
* had an investigational drug treatment within the previous 6 months; or
* pregnant and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Changes in net weight gain | Baseline, 3 week, 6 week, 9 week, 12 week
  Assessments will be conducted at baseline and once every three weeks thereafter.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) | Baseline, 3 week, 6 week, 9 week, 12 week
  Assessments will be conducted at baseline and once every three weeks thereafter.
Changes in waist circumference (WC) | Baseline, 3 week, 6 week, 9 week, 12 week
  Assessments will be conducted at baseline and once every three weeks thereafter.
Changes in blood pressure | Baseline, 6 week, 12 week
  Assessments will be conducted at baseline and once every six weeks thereafter.
Changes in triglycerides (TG) | Baseline, 12 week
  Triglycerides (TG) level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in total cholesterol | Baseline, 12 week
  Total cholesterol level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in high-density lipoprotein (HDL) | Baseline, 12 week
  High-density lipoprotein (HDL) level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in low-density lipoprotein (LDL) | Baseline, 12 week
  Low-density lipoprotein (LDL) level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in fasting glucose | Baseline, 12 week
  Fasting glucose level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in glycated haemoglobin (HbA1c) | Baseline, 12 week
  Glycated haemoglobin (HbA1c) level will be determined from blood samples collected at baseline and 12 weeks. The collection of blood will be conducted between 08:00 and 09:00 after an overnight fast.
Changes in positive and Negative Syndrome Scale (PANSS) | Baseline, 6 week, 12 week
  The severity of psychotic symptoms will be also assessed using the Positive and Negative Syndrome Scale (PANSS). Assessments will be conducted at baseline and once every six weeks thereafter.
Changes in extrapyramidal Symptom Rating Scale (ESRS) | Baseline, 6 week, 12 week
  The Extrapyramidal Symptom Rating Scale (ESRS) will be used to evaluate antipsychotic-induced movement symptoms. Assessments will be conducted at baseline and once every six weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin ZHANG, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- Castle Peak Hospital - The Department of General Adult Psychiatry, Tuenmen, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kane JM. Pharmacologic treatment of schizophrenia. Biol Psychiatry. 1999 Nov 15;46(10):1396-408. doi: 10.1016/s0006-3223(99)00059-1. PMID 10578454
- [Background] Bressington DT, Mui J, Cheung EF, Petch J, Clark AB, Gray R. The prevalence of metabolic syndrome amongst patients with severe mental illness in the community in Hong Kong--a cross sectional study. BMC Psychiatry. 2013 Mar 18;13:87. doi: 10.1186/1471-244X-13-87. PMID 23506322
- [Background] Pirillo A, Catapano AL. Berberine, a plant alkaloid with lipid- and glucose-lowering properties: From in vitro evidence to clinical studies. Atherosclerosis. 2015 Dec;243(2):449-61. doi: 10.1016/j.atherosclerosis.2015.09.032. Epub 2015 Sep 30. PMID 26520899
- [Background] Lan J, Zhao Y, Dong F, Yan Z, Zheng W, Fan J, Sun G. Meta-analysis of the effect and safety of berberine in the treatment of type 2 diabetes mellitus, hyperlipemia and hypertension. J Ethnopharmacol. 2015 Feb 23;161:69-81. doi: 10.1016/j.jep.2014.09.049. Epub 2014 Dec 10. PMID 25498346
- [Background] Hu Y, Young AJ, Ehli EA, Nowotny D, Davies PS, Droke EA, Soundy TJ, Davies GE. Metformin and berberine prevent olanzapine-induced weight gain in rats. PLoS One. 2014 Mar 25;9(3):e93310. doi: 10.1371/journal.pone.0093310. eCollection 2014. PMID 24667776
- [Background] Kulkarni SK, Dhir A. On the mechanism of antidepressant-like action of berberine chloride. Eur J Pharmacol. 2008 Jul 28;589(1-3):163-72. doi: 10.1016/j.ejphar.2008.05.043. Epub 2008 Jun 3. PMID 18585703
- [Background] Peng WH, Wu CR, Chen CS, Chen CF, Leu ZC, Hsieh MT. Anxiolytic effect of berberine on exploratory activity of the mouse in two experimental anxiety models: interaction with drugs acting at 5-HT receptors. Life Sci. 2004 Oct 1;75(20):2451-62. doi: 10.1016/j.lfs.2004.04.032. PMID 15350820
- [Background] Kawano M, Takagi R, Kaneko A, Matsushita S. Berberine is a dopamine D1- and D2-like receptor antagonist and ameliorates experimentally induced colitis by suppressing innate and adaptive immune responses. J Neuroimmunol. 2015 Dec 15;289:43-55. doi: 10.1016/j.jneuroim.2015.10.001. Epub 2015 Oct 14. PMID 26616870
- [Background] Salehi S, Filtz TM. Berberine possesses muscarinic agonist-like properties in cultured rodent cardiomyocytes. Pharmacol Res. 2011 Apr;63(4):335-40. doi: 10.1016/j.phrs.2010.12.004. Epub 2010 Dec 17. PMID 21168503
- [Background] Harsing LG Jr, Lonart G, Vizi SE. Berbanes: search for novel alpha-2 adrenoceptor antagonists. Pol J Pharmacol Pharm. 1988 Nov-Dec;40(6):697-708. PMID 2908367
- [Background] Wang HH, Cai M, Wang HN, Chen YC, Zhang RG, Wang Y, McAlonan GM, Bai YH, Wu WJ, Guo L, Zhang YH, Tan QR, Zhang ZJ. An assessor-blinded, randomized comparison of efficacy and tolerability of switching from olanzapine to ziprasidone and the combination of both in schizophrenia spectrum disorders. J Psychiatr Res. 2017 Feb;85:59-65. doi: 10.1016/j.jpsychires.2016.11.002. Epub 2016 Nov 4. PMID 27837658
- [Background] Haffner SM, Miettinen H, Stern MP. The homeostasis model in the San Antonio Heart Study. Diabetes Care. 1997 Jul;20(7):1087-92. doi: 10.2337/diacare.20.7.1087. PMID 9203442
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Gharabawi GM, Bossie CA, Lasser RA, Turkoz I, Rodriguez S, Chouinard G. Abnormal Involuntary Movement Scale (AIMS) and Extrapyramidal Symptom Rating Scale (ESRS): cross-scale comparison in assessing tardive dyskinesia. Schizophr Res. 2005 Sep 15;77(2-3):119-28. doi: 10.1016/j.schres.2005.03.008. PMID 15913963